CLINICAL TRIAL: NCT06310603
Title: Determinants and Outcomes of High vs. Low Ultra-processed Feeding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-23-42
Record Dates: First submitted 2023-12-13; First posted 2024-03-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Processed Food Group (Experimental)
  Interventions: Other: Low-Processed Food Diet
- Typical Diet Group (No Intervention)

INTERVENTIONS:
Other: Low-Processed Food Diet — Participants that receive intervention will be instructed to eat a diet rich in unprocessed/minimally-processed foods, as described by the NOVA food classification system
  Arms: Low-Processed Food Group

SUMMARY:
The goal of this clinical trial is to learn about, test, and compare health outcomes of high vs. low-processed feeding. The main question[s] it aims to answer are:

• Does consuming a diet rich in unprocessed food improve various health outcomes? Participants will either be instructed to consume a diet rich in unprocessed food for 6 months, or consume their typical diet for 6 months. At various points in the study there will be metabolic health data collected.

If there is a comparison group: Researchers will compare the low-processed group to the typical diet group to see if there are improvements in metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* rural county resident
* not meeting physical activity guidelines for adults
* consuming a typical Western diet (rich in UPF)

Exclusion Criteria:

* chronic diseases
* tobacco, vape, or illicit drug use
* overly active
* already on a restrictive diet (e.g., keto, intermittent fasting)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-09 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 1 year
  Using a standard scale, body weight in kg will be assessed
Body Composition | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), body composition will be assessed
Fat Mass Percentage | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), fat mass percentage will be assessed
Fat-Free Mass Percentage | 1 year
  Using Dual-energy X-ray absorptiometry(DXA), fat-free mass will be assessed

SECONDARY OUTCOMES:
Triglyceride Levels | 1 year
  Blood draw followed by a Piccolo scan will analyze Triglyceride levels in the blood
Glucose Levels | 1 year
  Blood draw followed by a Piccolo scan will analyze glucose in the blood
Cholesterol Levels | 1 year
  Blood draw followed by a Piccolo scan will analyze glucose in the blood
HDL | 1 year
  Blood draw followed by a Piccolo scan will analyze HDL in the blood
LDL | 1 year
  Piccolo scan will analyze LDL in the blood
Alanine transaminase (ALT) | 1 year
  Blood draw followed by a Piccolo scan will analyze ALT in the blood
Aspartate transaminase (AST) | 1 year
  Blood draw followed by a Piccolo scan will analyze AST in the blood

OTHER OUTCOMES:
Energy Intake | 1 year
  3-Day Food Logs will record caloric intake at various points
Energy Expenditure | 1 year
  Resting Metabolic Rate will be used to find resting energy expenditure and an accelerometer will measure expended energy through fitness, combined these will show energy expenditure
Gut Microbiome Collection | 1 year
  Stool kits administered for fecal collection will be used for gut microbiome collection

CONTACTS AND LOCATIONS:
Overall Officials: Sam Emerson, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Laboratory for Applied Nutrition and Exercise Science (LANES), Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided